CLINICAL TRIAL: NCT01448330
Title: A Sequence-randomized, Open-label, Single Dose, Crossover Study to Evaluate Pharmacokinetics and Safety After Oral Administration of Clopidogrel and Aspirin in Free Combination and Fixed-dose Combination as HCP0911 in Healthy Male Volunteers
Brief Title: A Bioequivalence Study Comparing Clopidogrel/Aspirin Combination Tablet With Coadministration of Clopidogrel and Aspirin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-CPAS-101
Record Dates: First submitted 2011-09-27; First posted 2011-10-07 (Estimated); Last update posted 2011-12-30 (Estimated); Status verified 2011-09

CONDITIONS: Healthy
Keywords: clopidogrel; aspinin; combination
MeSH Terms: interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HCP0911 (Experimental): clopidogrel/aspirin combination tablet
  Interventions: Drug: HCP0911 / clopidogrel, aspirin
- clopidorel and aspirin (Active Comparator): coadministration of clopidogrel and aspirin
  Interventions: Drug: HCP0911 / clopidogrel, aspirin

INTERVENTIONS:
Drug: HCP0911 / clopidogrel, aspirin — combination tablet vs coadministration

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics and safety after oral administration of clopidogrel and aspirin in free combination as HCP0911.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 55
* Signed informed consent

Exclusion Criteria:

* Has a history of hypersensitivity to IP ingredients
* Hypotension or hypertension
* Has a history of acute infection within 14days of screening

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Cmax | 0-24 hrs
AUC | 0-24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Jae-wook Ko, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea

REFERENCES:
- [Derived] Jung JA, Kim TE, Kim JR, Kim MJ, Huh W, Park KM, Lee SY, Ko JW. The pharmacokinetics and safety of a fixed-dose combination of acetylsalicylic acid and clopidogrel compared with the concurrent administration of acetylsalicylic acid and clopidogrel in healthy subjects: a randomized, open-label, 2-sequence, 2-period, single-dose crossover study. Clin Ther. 2013 Jul;35(7):985-94. doi: 10.1016/j.clinthera.2013.05.015. PMID 23870608